CLINICAL TRIAL: NCT06954740
Title: Clinical Study to Evaluate the Efficacy and Safety of Mesenchymal Stromal Cells (Amimestrocel ) in Patients With Acute Kidney Injury
Acronym: MSC-AKI-001
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiangmei, Principal Investigator, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2025-167; S2025-167 (Other: Ethics Committee of Chinese PLA General Hospital)
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Acute Kidney Injury
Keywords: mesenchymal stromal cells (MSCs); acute kidney injury(AKI)
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amimestrocel (Experimental): In experimental group,patients receive standard treatment and Amimestrocel is administered via Intravenous infusion on day 1, 4, 8,15.
  Interventions: Drug: Amimestrocel

INTERVENTIONS:
Drug: Amimestrocel — Amimestrocel will be administered at a target dose of 1×10E6 MSCs/kg body weight on day 1, 4, 8, 15.

SUMMARY:
This trial is to evaluate the efficacy and safety of Amimestrocel (human umbilical cord mesenchymal stromal cells) in the treatment of AKI patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years old; gender is not restricted.
2. According to the 2023 KDIGO diagnostic criteria for acute kidney injury (AKI), including those that occur during the course of the disease in various patients with chronic kidney disease (CKD), AKI can be diagnosed if any of the following conditions is met:

   ① The serum creatinine level increases by ≥ 26.5 μmol/L within 48 hours;

   ② The serum creatinine level increases by more than 1.5 times or higher than the baseline value within 7 days;

   ③ The urine output decreases (< 0.5 mL/kg/h) and persists for more than 6 hours; The baseline value of serum creatinine: The lowest creatinine value obtained in the outpatient department or ward within 3 months, and the longest time limit is the creatinine value within 1 year. If there is no such value, the serum creatinine can be estimated using the MDRD equation under the assumption that the baseline eGFR is 75 ml/min/1.73m².
3. .Ability to give informed consent.

Exclusion Criteria:

1. Post-renal AKI.
2. Acute kidney injury caused by glomerular diseases such as rapidly progressive glomerulonephritis, lupus nephritis, anti-neutrophil cytoplasmic antibody-associated nephritis, anti-glomerular basement membrane antibody-mediated nephritis, vasculitis, cryoglobulinemia, thrombotic microangiopathy, etc.
3. Hemodynamic instability.
4. Severe cardiovascular diseases.
5. Severe pulmonary dysfunction.
6. A history of intracerebral hemorrhage or cerebral infarction within the past six months.
7. Subjects with abnormal laboratory indicators: AST or ALT > 5 × upper limit of normal value (ULN); total bilirubin > 3 × ULN; white blood cell count < 2000/μL (2 × 10⁹/L), hemoglobin < 6 g/dL (60 g/L), neutrophils < 1000/μL (1 × 10⁹/L), platelets < 50000/μL (50 × 10⁹/L).
8. Uncontrollable infection.
9. Patients with active hepatitis B or hepatitis C virus infection, active tuberculosis, severe immunodeficiency diseases, human immunodeficiency virus (HIV) infection, etc.
10. Received systemic immunosuppressants or glucocorticoid treatment for more than one week within 30 days before enrollment.
11. Have received hemodialysis or peritoneal dialysis treatment.
12. Have a history of hematopoietic stem cell transplantation or solid organ transplantation.
13. Patients with a history of malignant tumor within the past 5 years.
14. Life expectancy is less than 1 month.
15. Those with a known history of severe allergy to component blood or blood products, or those with a history of allergy to heterologous proteins.
16. Lactating women, or female patients who have a pregnancy plan or an egg donation plan from the start of the study to the follow-up period, and male patients (or their partners) who have a fertility plan or a sperm donation plan from the start of the study to the follow-up period and are unwilling to take contraceptive measures.
17. Patients who participated in other interventional clinical trials within 1 month before enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
serum creatinine | Change from baseline at 28 days

SECONDARY OUTCOMES:
serum creatinine | Change from baseline at 8,15,21 days, and 2, 3 months.
Stage of AKI | Change from baseline at 8, 15, 21, 28 days, and 2, 3 months.
  Evaluate the staging of Acute Kidney Injury (AKI) according to KDIGO guidelines.
proportion of study participants with Renal Replacement Therapy(RRT) | proportion of study participants with RRT at 4, 8, 12 weeks and 12, 24 months
APACHE II or APACHE III | Change from baseline at 8, 15, 21, 28 days, 2, 3,12, 24 months
SOFA | Change from baseline at 8, 15, 21, 28 days, 2, 3,12, 24 months
  Sequential Organ Failure Assessment Score
all-cause mortality ratio | All-cause mortality ratio at 28 days
Mechanism exploration | Change from baseline at 8, 15, 28 days, 3 months.
  Explore the mechanism through blood tests（Serum/plasma concentrations (pg/ml) of biomarkers of inflammation. Proportion/total number of circulating T cells, B cells, NK cells, etc ） and urine tests(mRNA, miRNA, etc)
Adverse Event and Serious Adverse Event | Within 12 weeks after received Amimestrocel
secondary malignant disease | Within 24 months after received Amimestrocel
  Number of Participants with secondary malignant disease

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Beijing hospital, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Capital Medical University Affiliated Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Medical Center, Tsinghua University, Beijing, Beijing Municipality